CLINICAL TRIAL: NCT04691635
Title: MotOr, cogniTIVe and Imaging charactErization of Progressive Supranuclear Palsy Phenotypes: a Longitudinal Prospective Study Looking for Biomarkers
Brief Title: The MOTIVE-PSP Initiative (Progressive Supranuclear Palsy)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Salerno (Other)
Collaborators: Azienda Ospedaliera di Padova (Other); Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Marina Picillo, Doctor, University of Salerno
Other Study IDs: CEMAND-2020-02
Record Dates: First submitted 2020-12-28; First posted 2020-12-31 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Progressive Supranuclear Palsy
MeSH Terms: conditions — Supranuclear Palsy, Progressive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Patients with Progressive Supranuclear Palsy
  Interventions: Other: evaluation of movements with sensors
- Group 2: Patients with Parkinson's disease
  Interventions: Other: evaluation of movements with sensors
- Group 3: Healthy controls
  Interventions: Other: evaluation of movements with sensors

INTERVENTIONS:
Other: evaluation of movements with sensors — evaluation of movements with sensors

SUMMARY:
Progressive Supranuclear Palsy (PSP) is a rapidly progressive neurodegenerative disease characterized by falls and oculomotor disturbances. Several clinical trials are currently evaluating the efficacy of new pharmacological compounds in slowing disease progression. Yet, both early diagnosis and evaluation of disease progression remain challenging.

Study aims include verifying if specific motor, cognitive, language, cerebrospinal fluid and imaging assessments represent reliable biomarkers of PSP diagnosis, phenotypization and progression over 1-year follow up. Motor evaluation will include recordings from wearable sensors.

Expected results include 1) improvement of PSP diagnosis and phenotypization; 2)improvement of evaluation of disease progression in the context of clinical trial; 3)enhancement of strategies to prevent falls and fractures in such patients leading, in turn, to significant cost savings for the National Health System.

DETAILED DESCRIPTION:
Hyphotesis and Significance:

1)Cross-sectional phase:verify if specific motor, cognitive, language, cerebrospinal fluid (CSF) and imaging assessments represent reliable biomarkers of diagnosis in PSP in the earliest stages of disease compared to Parkinson's disease (PD) and healthy controls (HC) and are able characterize the different PSP clinical phenotype 2)12-month longitudinal phase:verify if specific motor, cognitive, language, CSF and imaging assessments represent reliable biomarkers of disease progression also according to the clinical phenotype

Preliminary Data:

Cross-sectional data suggest that current motor, cognitive, language and imaging assessments may be useful in supporting the diagnosis of PSP compared to PD and HC, but not in characterizing the PSP clinical phenotypes. No robust data on wearable sensors and CSF biomarkers is available.

Longitudinal data on such biomarkers are lacking. As for cognition, preliminary data suggest that the Repeatable Battery for the assessment of neuropsychological status (RBANS) may evaluate cognitive trajectories in PSP with Richardson's syndrome.

Specific Aim 1:

Determine the feasibility, validity and reliability of application of digital biomarkers in PSP. Specifically if clinic-based wearable sensors and smartphone-based remote assessments can (1) support early clinical diagnosis and phenotyping of PSP patients compared to PD and HC and (2) evaluate disease trajectories in the whole cohort of PSP patients and discrete phenotypes compared to standard rating scales.

For both points the hypothesis is that both clinic-based and smartphone-based wearable sensors outperform standard rating scales.

Specific aim 2:

Verify if cognitive, language and behavioral testing can (1) support early clinical diagnosis and phenotyping of PSP patients compared to PD and HC and (2) evaluate disease trajectories in the whole cohort of PSP patients and discrete phenotypes.

For point (1) the hypothesis is that cognitive, language and behavioral testing support early diagnosis and phenotyping in the earliest stages compared to PD and HC. For point (2) the hypothesis is that cognitive, language and behavioral testing are able to evaluate disease progression in the whole cohort of PSP patients and discrete phenotypes.

Specific aim 3:

Verify if single parameter and multiparameter magnetic resonance imaging (MRI) imaging assessments can (1) support early clinical diagnosis and phenotyping of PSP patients compared to PD and HC and (2) evaluate disease trajectories in the whole cohort of PSP patients and discrete phenotypes.

Experimental design aim 1 includes a cross-sectional phase with enrollment of 3 groups of subjects (PSP, PD and HC).

During the baseline evaluation each enrolled subject will perform:1) a clinic-based standardized protocol for assessment of gait with wearable inertial sensors to specifically monitor quality of gait and balance using a wide range of measures from the upper and lower body (APDM Mobility Lab system) ;2) home-based monitoring with smartphone of inertial measurement (balance and gait task) and voice recorded with microphone for at least 5 days;3) standard clinical rating scales including the PSP rating scale, the Natural History and Neuroprotection in Parkinson Plus Syndromes, Movement Disorder Society Unified Parkinson's disease rating scale part III, Falls diary to be filled during the 5-day home based monitoring. Caregivers will be asked to actively support patients for the home- smartphone-based digital biomarkers measurements.

Furthermore, at baseline only PSP patients will be asked to perform lumbar puncture to collect CSF and measure total-tau, phosphorylated tau, Beta-amyloid 42, neurofilament light and heavy chain. A 12-month longitudinal phase will follow only for PSP patients.

During both cross-sectional and longitudinal phases (every 3 months), only patients enrolled at Unit 1 will also perform a gait analysis assessment with a traditional opto-kinematic, hospital-based gait analysis system (Qualisys®, Sandvälen, Sweden).

Experimental design aim 2 includes a cross-sectional phase with enrollment of 3 groups of subjects (PSP, PD and HC).

During the baseline evaluation each enrolled subject will perform:1) the RBANS; 2)standard cognitive assessment currently used by part of the research team to evaluate cognitive abilities in PSP patients as detailed elsewhere; 3) functional autonomy will be evaluated with the Instrumental Activities of Daily Life, while depression and apathy with the Beck Depression Inventory II and Apathy Evaluation Scale, respectively; 4) other neuropsychiatric symptoms will be explored with the Neuropsychiatric Inventory; 5) language abilities will be explored with the Screening for Aphasia in NeuroDegeneration (SAND) battery.

A 12-month longitudinal phase will follow only for PSP patients.

Experimental design aim 3 includes a cross-sectional phase with enrollment of 3 groups of subjects (PSP, PD and HC).

During the baseline evaluation each enrolled subject will undergo a multimodal 3T MRI. The MRI protocol will include conventional sequences for morphometric measures (ie, the superior cerebellar peduncles, the middle cerebellar peduncles, the MR Parkinsonism index, the midbrain-pons area ratio; a 3D Spoiled Gradient Recalled Echo (SPGR) and a 3D-GRE multi-echo susceptibility weighted (SWAN) images to obtain quantitative susceptibility mapping and ROI based measures in substantia nigra, basal ganglia thalamus, red nucleus and fronto-parietal cortex, a resting state functional MRI and an Arterial Spin Labeling sequence.

A 12-month longitudinal phase will follow only for PSP patients. Both single parameter and multiparameter (morphometric, iron based, functional, and perfusion) MRI approaches will be applied to validate the usefulness of imaging assessments in predicting both early PSP diagnosis and phenotyping as well as disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Progressive Supranuclear Palsy based on current available clinical criteria
* ability to walk for at least 5 steps

Exclusion Criteria:

* Comorbidities interfering with study assessments
* Significant MRI abnormalities as cerebrovascular diseases, tumors.

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Progressive Supranuclera palsy. Any phenotype of the disease will be included
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Progressive Supranuclear Palsy rating scale | 1-year follow up
  Progression of disease as assessed with the standard clinical scale rating (scoring 0-100, higher scores indicate worse scores) Progressive Supranuclear Palsy symptoms and signs

SECONDARY OUTCOMES:
Cognitive progression | 1-year follow up
  Evaluated with the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) scale score (scoring 0-100, higher scores indicate better scores)
Behavioral progression | 1-year follow up
  Behavioral symptoms as assessed with Neuropsychiatric Inventory scale (scoring 0-144, higher scores indicate worse scores)
MRI | 1-year follow up
  Progression of disease as assessed with MRI specific measures (the superior cerebellar peduncles, the middle cerebellar peduncles, the MR Parkinsonism index, the midbrain-pons area ratio; a 3D Spoiled Gradient Recalled Echo (SPGR) and a 3D-GRE multi-echo susceptibility weighted)
Gait speed | 1-year follow up
  Gait speed as assessed with motion sensors

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - AOU Padova, Padua
  - AOU Pisa, Pisa
  - AOU San Giovanni di Dio e Ruggi d'Aragona, Salerno

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with external researchers

REFERENCES:
- [Background] Picillo M, Abate F, Ponticorvo S, Tepedino MF, Erro R, Frosini D, Del Prete E, Cecchi P, Cosottini M, Ceravolo R, Salle GD, Salle FD, Esposito F, Pellecchia MT, Manara R, Barone P. Association of MRI Measures With Disease Severity and Progression in Progressive Supranuclear Palsy. Front Neurol. 2020 Nov 12;11:603161. doi: 10.3389/fneur.2020.603161. eCollection 2020. PMID 33281738
- [Background] Picillo M, Cuoco S, Carotenuto I, Abate F, Erro R, Volpe G, Pellecchia MT, Catricala E, Cappa S, Barone P. Clinical use of SAND battery to evaluate language in patients with Progressive Supranuclear Palsy. PLoS One. 2019 Oct 11;14(10):e0223621. doi: 10.1371/journal.pone.0223621. eCollection 2019. PMID 31603934
- [Background] Picillo M, Tepedino MF, Abate F, Erro R, Ponticorvo S, Tartaglione S, Volpe G, Frosini D, Cecchi P, Cosottini M, Ceravolo R, Esposito F, Pellecchia MT, Barone P, Manara R. Midbrain MRI assessments in progressive supranuclear palsy subtypes. J Neurol Neurosurg Psychiatry. 2020 Jan;91(1):98-103. doi: 10.1136/jnnp-2019-321354. Epub 2019 Sep 16. PMID 31527182
- [Background] Picillo M, Cuoco S, Amboni M, Bonifacio FP, Bruschi F, Carotenuto I, De Micco R, De Rosa A, Del Prete E, Di Biasio F, Elifani F, Erro R, Fabbri M, Falla M, Franco G, Frosini D, Galantucci S, Lazzeri G, Magistrelli L, Malaguti MC, Milner AV, Minafra B, Olivola E, Pilotto A, Rascuna C, Rizzetti MC, Schirinzi T, Borroni B, Ceravolo R, Di Fonzo A, Marchese R, Mercuri NB, Modugno N, Nicoletti A, Padovani A, Santangelo G, Stefani A, Tessitore A, Volonte MA, Zangaglia R, Zappia M, Zibetti M, Barone P. Validation of the Italian version of the PSP Quality of Life questionnaire. Neurol Sci. 2019 Dec;40(12):2587-2594. doi: 10.1007/s10072-019-04010-2. Epub 2019 Jul 26. PMID 31350659
- [Background] Picillo M, Cuoco S, Amboni M, Bonifacio FP, Bruno A, Bruschi F, Cappiello A, De Micco R, De Rosa A, Di Biasio F, Elifani F, Erro R, Fabbri M, Falla M, Franco G, Frosini D, Galantucci S, Lazzeri G, Magistrelli L, Malaguti MC, Milner AV, Minafra B, Olivola E, Pilotto A, Rascuna C, Rizzetti MC, Schirinzi T, Borroni B, Ceravolo R, Di Fonzo A, Lopiano L, Marchese R, Mercuri NB, Modugno N, Nicoletti A, Padovani A, Santangelo G, Stefani A, Tessitore A, Volonte MA, Zangaglia R, Zappia M, Barone P. Validation of the Italian version of carers' quality-of-life questionnaire for parkinsonism (PQoL Carer) in progressive supranuclear palsy. Neurol Sci. 2019 Oct;40(10):2163-2169. doi: 10.1007/s10072-019-03944-x. Epub 2019 Jun 12. PMID 31190253
- [Background] Picillo M, Cuoco S, Tepedino MF, Cappiello A, Volpe G, Erro R, Santangelo G, Pellecchia MT, Barone P; PSP Salerno study group. Motor, cognitive and behavioral differences in MDS PSP phenotypes. J Neurol. 2019 Jul;266(7):1727-1735. doi: 10.1007/s00415-019-09324-x. Epub 2019 Apr 15. PMID 30989369
- [Background] Picillo M, Erro R, Cuoco S, Tepedino MF, Manara R, Pellecchia MT, Barone P; PSP Salerno Study Group. MDS PSP criteria in real-life clinical setting: Motor and cognitive characterization of subtypes. Mov Disord. 2018 Aug;33(8):1361-1365. doi: 10.1002/mds.27408. Epub 2018 Jul 8. No abstract available. PMID 29984518